CLINICAL TRIAL: NCT00635674
Title: Effects of CPAP on Cardiovascular Risk Profile in Patients With Severe Obstructive Sleep Apnea and Metabolic Syndrome
Brief Title: Effects of CPAP on Cardiovascular Risk in Obstructive Sleep Apnea (OSA) and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Ruzena Tkacova, MD, PhD, Professor of Medicine, Medical Faculty, PJ Safarik University and L. Pasteur Teaching Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSAMSCPAP
Record Dates: First submitted 2008-02-25; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Obstructive Sleep Apnea; Metabolic Syndrome
Keywords: sleep apnea; risk factors; continuous positive airway pressure; insulin resistance; metabolic syndrome; compliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Metabolic Syndrome; Sleep Apnea Syndromes; Insulin Resistance; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I - compliant (Experimental): CPAP use for more than 4 hr/night
  Interventions: Device: CPAP device - REMstar Plus, Respironics, Murrysville, USA
- Group 2-noncompliant (Active Comparator): CPAP for less than 4 hr/night
  Interventions: Device: CPAP device - REMstar Plus, Respironics, Murrysville, USA

INTERVENTIONS:
Device: CPAP device - REMstar Plus, Respironics, Murrysville, USA — continuous positive airway pressure device with heated humidification
  Other Names: REMstar Plus, Respironics, Murrysville, Pennsylvania, USA

SUMMARY:
The increased risk of atherosclerotic morbidity and mortality in patients with obstructive sleep apnea (OSA) has been linked to arterial hypertension, insulin resistance, systemic inflammation, and oxidative stress in previous studies.

We aimed to determine the effects of 8-weeks therapy with continuous positive airway pressure (CPAP) on glucose and lipid profile, systemic inflammation, oxidative stress, and the global cardiovascular disease (CVD) risk in patients with severe OSA and metabolic syndrome.

DETAILED DESCRIPTION:
Patients with obstructive sleep apnea (OSA) are at increased risk of atherosclerotic morbidity and mortality.OSA is associated with the development and/or worsening of arterial hypertension, a traditional risk factor of atherosclerosis.Moreover, OSA has been linked to novel factors related to atherogenesis - metabolic syndrome,systemic inflammation,6 and oxidative stress.

Numerous studies have selectively examined the effects of continuous positive airway pressure (CPAP) ventilation, the primary treatment for OSA, on the traditional and novel risk factors of atherosclerosis. A recent metaanalysis of 16 randomized trials indicated that CPAP decreases blood pressure in patients with OSA.9 Furthermore, reductions in serum total cholesterol, C-reactive protein (CRP), tumor necrosis factor-alpha (TNF-alpha), interleukin (IL)-6 and IL-8 were demonstrated after effective CPAP therapy.In addition, CPAP was shown to reduce systemic oxidative stress.Improvements in insulin sensitivity have been reported in some,but not in all studies. Importantly, substantial evidence links the effects of CPAP to compliance with this treatment.

Most observational studies examined the effects of CPAP across a broad-range of OSA severity, and have included patients with and without the metabolic syndrome. Up to now, no study analyzed the effects of CPAP on glucose and lipid metabolism, systemic inflammation, oxidative stress, and the global cardiovascular disease (CVD) risk within the same cohort of subjects with severe OSA and concurrent metabolic syndrome. Importantly, the metabolic syndrome exacerbates CVD risk over and above that attributable to OSA alone. Therefore, reduction of CVD risk in patients with OSA and concurrent metabolic syndrome is of paramount importance.

The primary purpose of the present study was to determine, in patients with severe OSA and metabolic syndrome compliant to CPAP, the effects of 8-weeks therapy on the glucose and lipid profile, systemic inflammation, oxidative stress, and on the global CVD risk. The secondary goal was to analyze factors related to compliance with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* severe OSA (more than 30 obstructive apneas or hypopneas per hour of sleep and excessive daytime sleepiness)
* metabolic syndrome

Exclusion Criteria:

* endocrine or metabolic disorders other than metabolic syndrome
* history of myocardial infarction, angina or stroke
* inflammatory or other chronic disease
* respiratory disorder other than OSA
* neurological lesions
* regular use of sedative medication or alcohol

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease risk profile (as assessed using the multivariable risk factor algorithm) | 8 weeks therapy with Continuous positive airway pressure

SECONDARY OUTCOMES:
insulin sensitivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruzena Tkacova, MD,PhD, Principal Investigator — Head, Department of Respiratory Medicine, Medical Faculty PJ SAfarik University and L Pasteur Teaching Hospital
Locations (1):
- Medical Faculty, PJ Safarik University, Košice, Slovakia, Slovakia

REFERENCES:
- [Derived] Dorkova Z, Petrasova D, Molcanyiova A, Popovnakova M, Tkacova R. Effects of continuous positive airway pressure on cardiovascular risk profile in patients with severe obstructive sleep apnea and metabolic syndrome. Chest. 2008 Oct;134(4):686-692. doi: 10.1378/chest.08-0556. Epub 2008 Jul 14. PMID 18625666